CLINICAL TRIAL: NCT02037984
Title: A Phase I-II, Randomized, Double-Blind, Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Healthy Adults and Infants
Brief Title: Safety, Tolerability and Immunogenicity of V114 in Healthy Adults and Infants (V114-004)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-004
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Streptococcus Pneumoniae Infection; Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Adult V114: 1x:1x:1x (Experimental): Adults receive a single vaccination on Day 1.
  Interventions: Biological: V114 1x:1x:1x
- Adult V114: 2x:2x:2x (Experimental): Adults receive a single vaccination on Day 1.
  Interventions: Biological: V114 2x:2x:2x
- Infant V114: 1x:1x:1x (Experimental): Infants receive 4 total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 1x:1x:1x
- Infant V114: 2x:1x:2x (Experimental): Infants receive 4 total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 2x:1x:2x
- Infant V114: 2x:2x:2x (Experimental): Infants receive 4 total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 2x:2x:2x
- Infant V114: 0.5x:0.5x:2x (Experimental): Infants receive 4 total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 0.5x:0.5x:2x
- Infant V114: 1x:1x:2x (Experimental): Infants receive 4 total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 1x:1x:2x
- Infant Prevnar 13® (Active Comparator): Infants receive 4 total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: Prevnar 13®

INTERVENTIONS:
Biological: Prevnar 13® — Pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 µg each), and 6B (4.4 µg) in each 0.5 mL dose.
  Arms: Infant Prevnar 13®
Biological: V114 1x:1x:1x — V114 1x:1x:1x contains 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 125 µg of Aluminum Phosphate Adjuvant (APA).
  Arms: Adult V114: 1x:1x:1x; Infant V114: 1x:1x:1x
Biological: V114 2x:2x:2x — V114 2x:2x:2x contains 4.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 µg of APA.
  Arms: Adult V114: 2x:2x:2x; Infant V114: 2x:2x:2x
Biological: V114 2x:1x:2x — V114 2x:1x:2x contains 4.0 μg of polysaccharide serotypes 6A, 18C, 19A, 19F, and 23F; 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 7F, 9V, 14, 22F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 µg of APA.
  Arms: Infant V114: 2x:1x:2x
Biological: V114 1x:1x:2x — V114 1x:1x:2x contains 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 250 µg of APA.
  Arms: Infant V114: 1x:1x:2x
Biological: V114 0.5x:0.5x:2x — V114 0.5x:0.5x:2x contains 1.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 2.0 μg of polysaccharide serotype 6B; and 250 µg of APA.
  Arms: Infant V114: 0.5x:0.5x:2x

SUMMARY:
This study is designed to assess the safety, tolerability, and immunogenicity of 5 different formulations of V114 in healthy adults and infants. Adults only will be enrolled in Period 1 and infants only will be enrolled in Period 2; Period 1 will complete prior to the start of Period 2.

ELIGIBILITY:
Inclusion Criteria

Infants:

- Healthy and able to attend all scheduled visits.

Adults:

- Highly unlikely to conceive from vaccination to 6 weeks after administration of the vaccine.

Exclusion Criteria

Infants and Adults:

* Prior administration of any pneumococcal vaccine, any non-live vaccine within 14 days, or any live vaccine within 30 days.
* History of invasive pneumococcal disease.
* Known hypersensitivity to any vaccine component.
* Received systemic corticosteroids within 14 days of first vaccination.
* Known or suspected impairment of immune function.
* Febrile illness within 72 hours before vaccination.
* Received blood transfusion or blood products within 30 days. Infants
* Mother has documented human immunodeficiency virus or is hepatitis B surface antigen positive.
* Has asplenia or failure to thrive.

Adults:

- Is breastfeeding.

Ages: 6 Weeks to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 341 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rupp R, Hurley D, Grayson S, Li J, Nolan K, McFetridge RD, Hartzel J, Abeygunawardana C, Winters M, Pujar H, Benner P, Musey L. A dose ranging study of 2 different formulations of 15-valent pneumococcal conjugate vaccine (PCV15) in healthy infants. Hum Vaccin Immunother. 2019;15(3):549-559. doi: 10.1080/21645515.2019.1568159. Epub 2019 Feb 15. PMID 30689507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults and infants were recruited and enrolled at 26 study sites in the United States. Each of the adult participants completed the study prior to enrollment of the infant participants.
Groups:
- Adult V114: 1x:1x:1x: On Day 1, adults receive a single vaccination of V114 1x:1x:1x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 125 µg of Aluminum Phosphate Adjuvant [APA]).
- Adult V114: 2x.2x.2x: On Day 1, adults receive a single vaccination of V114 2x:2x:2x (containing 4.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 µg of APA).
- Infant V114: 1x:1x:1x: Infants receive 4 total V114: 1x:1x:1x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 125 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant V114: 2x:1x:2x: Infants receive 4 total V114: 2x:1x:2x (containing 4.0 μg of polysaccharide serotypes 6A, 18C, 19A, 19F, and 23F; 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 7F, 9V, 14, 22F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant V114: 2x:2x:2x: Infants receive 4 total V114: 2x:2x:2x (containing 4.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant V114: 0.5x:0.5x:2x: Infants receive 4 total V114 0.5x:0.5x:2x (containing 1.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 2.0 μg of polysaccharide serotype 6B; and 250 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant V114: 1x:1x:2x: Infants receive 4 total V114 1x:1x:2x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 250 µg of APA) total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant Prevnar 13®: Infants receive 4 total Prevnar 13® (containing 2.2 µg of pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, and 23F; and 4.4 µg of serotype 6B) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
Period: Overall Study
Arm/Group | Adult V114: 1x:1x:1x | Adult V114: 2x.2x.2x | Infant V114: 1x:1x:1x | Infant V114: 2x:1x:2x | Infant V114: 2x:2x:2x | Infant V114: 0.5x:0.5x:2x | Infant V114: 1x:1x:2x | Infant Prevnar 13®
Started (Randomized) | 20 | 20 | 50 | 51 | 50 | 49 | 50 | 51
Completed | 19 | 20 | 38 | 30 | 38 | 37 | 33 | 39
Not Completed | 1 | 0 | 12 | 21 | 12 | 12 | 17 | 12
Not completed — Lack of Efficacy | 0 | 0 | 3 | 10 | 2 | 2 | 4 | 3
Not completed — Lost to Follow-up | 1 | 0 | 3 | 5 | 2 | 2 | 2 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Technical Problems | 0 | 0 | 3 | 3 | 2 | 3 | 4 | 2
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 3 | 2 | 5 | 1 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants are included. One participant in the Infant V114: 0.5x:0.5x:2x arm was enrolled and randomized but did not receive any study treatment.
Groups:
- Adult V114: 1x:1x:1x: On Day 1, adults receive a single vaccination of V114 1x:1x:1x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 125 µg of APA).
- Total: Total of all reporting groups
Arm/Group | Adult V114: 1x:1x:1x | Adult V114: 2x.2x.2x | Infant V114: 1x:1x:1x | Infant V114: 2x:1x:2x | Infant V114: 2x:2x:2x | Infant V114: 0.5x:0.5x:2x | Infant V114: 1x:1x:2x | Infant Prevnar 13® | Total
Number analyzed (Participants) | 20 | 20 | 50 | 51 | 50 | 48 | 50 | 51 | 340
Age, Continuous [Mean (Standard Deviation); unit: Years] — Mean (SD) age in years is shown for adults. Population: Adult participants only are included.
  Years
    number analyzed (Participants) | 20 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 40
    (all) | 31.3 (8.9) | 31.6 (8.1) |  |  |  |  |  |  | 31.4 (8.4)
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Mean (SD) age in weeks is shown for infants. Population: Infant participants only are included.
  Weeks
    number analyzed (Participants) | 0 | 0 | 50 | 51 | 50 | 48 | 50 | 51 | 300
    (all) |  |  | 8.9 (1.4) | 8.7 (1.2) | 8.9 (1.3) | 8.5 (1.5) | 8.6 (1.0) | 8.4 (1.0) | 8.7 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 30 | 26 | 23 | 18 | 28 | 30 | 182
  Male | 5 | 8 | 20 | 25 | 27 | 30 | 22 | 21 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Black or African American | 3 | 4 | 3 | 5 | 4 | 8 | 2 | 4 | 33
  White | 15 | 15 | 42 | 44 | 41 | 35 | 46 | 42 | 280
  More than one race | 0 | 1 | 4 | 2 | 4 | 5 | 2 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adult Participants Experiencing ≥1 Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 14 days
Population: Adult participants who received V114 are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Adult V114: 1x:1x:1x | Adult V114: 2x.2x.2x
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 100.0 | 100.0

2. Primary Outcome: Percentage of Adult Participants Discontinuing From Study Treatment Due to an Adverse Event (AE)
Description: as for outcome 1
Time Frame: Up to 14 days
Population: Adult participants who received V114 are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Adult V114: 1x:1x:1x | Adult V114: 2x.2x.2x
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 0.0 | 0.0

3. Primary Outcome: Percentage of Infant Participants Experiencing ≥1 Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. For infants, AEs were monitored for up to 14 days following each vaccination.
Time Frame: Up to 14 days after the 4th vaccination (approximately 12.5 to 15.5 months of age)
Population: Infant participants who received V114 are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infant V114: 1x:1x:1x | Infant V114: 2x:1x:2x | Infant V114: 2x:2x:2x | Infant V114: 0.5x:0.5x:2x | Infant V114: 1x:1x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51 | 50 | 48 | 50 | 51
Percentage of Participants | 98.0 | 100.0 | 96.0 | 97.9 | 98.0 | 98.0

4. Primary Outcome: Percentage of Infant Participants Discontinuing From Study Treatment Due to an Adverse Event (AE)
Description: as for outcome 3
Time Frame: Up to 14 days after the 4th vaccination (approximately 12.5 to 15.5 months of age)
Population: Infant participants who received V114 are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infant V114: 1x:1x:1x | Infant V114: 2x:1x:2x | Infant V114: 2x:2x:2x | Infant V114: 0.5x:0.5x:2x | Infant V114: 1x:1x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51 | 50 | 48 | 50 | 51
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

5. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibodies at 1 Month Postdose 3 (PD3) in Infants: V114 1x:1x:1x vs. Prevnar 13®
Description: The IgG antibody GMCs of each Prevnar 13®-type (PT) or non-Prevnar 13® type (non-PT) serotype at 1 month PD3 following V114 or Prevnar 13® treatment were determined with the pneumococcal electrochemiluminescence (Pn ECL) assay. Data reflect the GMC of each serotype.
Time Frame: Month 7 (1 month PD3)
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infant V114: 1x:1x:1x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51
µg/mL
  PT1: number analyzed (Participants) | 38 | 40
  PT1 | 1.20 [0.98 to 1.48] | 1.48 [1.20 to 1.83]
  PT3: number analyzed (Participants) | 38 | 40
  PT3 | 0.96 [0.75 to 1.22] | 0.43 [0.35 to 0.54]
  PT4: number analyzed (Participants) | 38 | 40
  PT4 | 1.33 [1.07 to 1.66] | 0.98 [0.78 to 1.22]
  PT5: number analyzed (Participants) | 38 | 40
  PT5 | 1.16 [0.88 to 1.53] | 1.63 [1.25 to 2.14]
  PT6A: number analyzed (Participants) | 38 | 39
  PT6A | 1.64 [1.04 to 2.61] | 2.75 [2.28 to 3.31]
  PT6B: number analyzed (Participants) | 38 | 40
  PT6B | 0.77 [0.45 to 1.32] | 2.24 [1.54 to 3.24]
  PT7F: number analyzed (Participants) | 38 | 40
  PT7F | 2.09 [1.65 to 2.64] | 2.90 [2.48 to 3.39]
  PT9V: number analyzed (Participants) | 38 | 40
  PT9V | 1.00 [0.75 to 1.33] | 1.35 [1.05 to 1.74]
  PT14: number analyzed (Participants) | 38 | 40
  PT14 | 2.96 [1.95 to 4.48] | 5.01 [3.94 to 6.38]
  PT18C: number analyzed (Participants) | 38 | 40
  PT18C | 1.29 [1.05 to 1.60] | 1.41 [1.14 to 1.74]
  PT19A: number analyzed (Participants) | 38 | 40
  PT19A | 1.27 [0.99 to 1.62] | 1.45 [1.13 to 1.86]
  PT19F: number analyzed (Participants) | 38 | 40
  PT19F | 2.31 [1.75 to 3.04] | 1.89 [1.56 to 2.30]
  PT23F: number analyzed (Participants) | 38 | 40
  PT23F | 1.02 [0.75 to 1.40] | 1.13 [0.87 to 1.47]
  non-PT22F: number analyzed (Participants) | 38 | 40
  non-PT22F | 4.10 [3.04 to 5.53] | 0.06 [0.05 to 0.08]
  non-PT33F: number analyzed (Participants) | 38 | 40
  non-PT33F | 1.37 [0.84 to 2.22] | 0.06 [0.04 to 0.08]
Statistical Analysis 1: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT1 GMC Ratio (V114/Prevnar 13®); PT1 GMC Ratio = 0.81, 95% CI 2-sided [0.60 to 1.10]
Statistical Analysis 2: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT3 GMC Ratio (V114/Prevnar 13®); PT3 GMC Ratio = 2.22, 95% CI 2-sided [1.64 to 3.02]
Statistical Analysis 3: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT4 GMC Ratio (V114/Prevnar 13®); PT4 GMG Ratio = 1.37, 95% CI 2-sided [1.01 to 1.84]
Statistical Analysis 4: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT5 GMC Ratio (V114/Prevnar 13®); PT5 GMC Ratio = 0.71, 95% CI 2-sided [0.48 to 1.05]
Statistical Analysis 5: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT6A GMC Ratio (V114/Prevnar 13®); PT6A GMC Ratio = 0.60, 95% CI 2-sided [0.32 to 1.13]
Statistical Analysis 6: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT6B GMC Ratio (V114/Prevnar 13®); PT6B GMG Ratio = 0.34, 95% CI 2-sided [0.16 to 0.73]
Statistical Analysis 7: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT7F GMC Ratio (V114/Prevnar 13®); PT7F GMC Ratio = 0.72, 95% CI 2-sided [0.51 to 1.02]
Statistical Analysis 8: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT9V GMC Ratio (V114/Prevnar 13®); PT9V GMC Ratio = 0.74, 95% CI 2-sided [0.51 to 1.08]
Statistical Analysis 9: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT14 GMC Ratio (V114/Prevnar®); PT9V GMC Ratio = 0.59, 95% CI 2-sided [0.39 to 0.90]
Statistical Analysis 10: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT18C GMC Ratio (V114/Prevnar 13®); PT18C GMC Ratio = 0.92, 95% CI 2-sided [0.64 to 1.31]
Statistical Analysis 11: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT19A GMC Ratio (V114/Prevnar 13®); PT19A GMC Ratio = 0.88, 95% CI 2-sided [0.61 to 1.27]
Statistical Analysis 12: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT19F GMC Ratio (V114/Prevnar 13®); PT19F GMC Ratio = 1.22, 95% CI 2-sided [0.83 to 1.78]
Statistical Analysis 13: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT23F GMC Ratio (V114/Prevnar 13®); PT23F GMC Ratio = 0.91, 95% CI 2-sided [0.57 to 1.45]
Statistical Analysis 14: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — non-PT22F GMC Ratio (V114/Prevnar 13®); non-PT22F GMC Ratio = 67.50, 95% CI 2-sided [45.58 to 99.97]
Statistical Analysis 15: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — non-PT33F GMC Ratio (V114/Prevnar 13®); non-PT33F GMC Ratio = 23.90, 95% CI 2-sided [13.21 to 43.24]

6. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibodies at 1 Month Postdose 3 (PD3) in Infants: V114 2x:1x:2x vs. Prevnar 13®
Description: as for outcome 5
Time Frame: Month 7 (1 month PD3)
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Infant V114: 2x:1x:2x: Infants receive 4 total V114: 2x:1x:2x (containing 4.0 μg of polysaccharide serotypes 6A, 18C, 19A, 19F, and 23F; 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 7F, 9V, 14, 22F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 μg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
Arm/Group | Infant V114: 2x:1x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 51 | 51
µg/mL
  PT1: number analyzed (Participants) | 42 | 40
  PT1 | 0.77 [0.60 to 0.99] | 1.48 [1.20 to 1.83]
  PT3: number analyzed (Participants) | 42 | 40
  PT3 | 0.77 [0.60 to 0.99] | 0.43 [0.35 to 0.54]
  PT4: number analyzed (Participants) | 42 | 40
  PT4 | 0.85 [0.70 to 1.02] | 0.98 [0.78 to 1.22]
  PT5: number analyzed (Participants) | 42 | 40
  PT5 | 0.83 [0.70 to 1.02] | 1.63 [1.25 to 2.14]
  PT6A: number analyzed (Participants) | 42 | 39
  PT6A | 0.85 [0.49 to 1.48] | 2.75 [2.28 to 3.31]
  PT6B: number analyzed (Participants) | 42 | 40
  PT6B | 0.36 [0.19 to 0.69] | 2.24 [1.54 to 3.24]
  PT7F: number analyzed (Participants) | 42 | 40
  PT7F | 1.39 [1.10 to 1.77] | 2.90 [2.48 to 3.39]
  PT 9V: number analyzed (Participants) | 42 | 40
  PT 9V | 0.76 [0.58 to 1.00] | 1.35 [1.05 to 1.74]
  PT14: number analyzed (Participants) | 42 | 40
  PT14 | 3.20 [2.37 to 4.33] | 5.01 [3.94 to 6.38]
  PT18C: number analyzed (Participants) | 42 | 40
  PT18C | 1.20 [0.92 to 1.57] | 1.41 [1.14 to 1.74]
  PT19A: number analyzed (Participants) | 42 | 40
  PT19A | 0.96 [0.75 to 1.23] | 1.45 [1.13 to 1.86]
  PT19F: number analyzed (Participants) | 42 | 40
  PT19F | 2.10 [1.57 to 2.81] | 1.89 [1.56 to 2.30]
  PT23F: number analyzed (Participants) | 42 | 40
  PT23F | 0.76 [0.51 to 1.13] | 1.13 [0.87 to 1.47]
  non-PT22F: number analyzed (Participants) | 42 | 40
  non-PT22F | 2.71 [1.95 to 3.78] | 0.06 [0.05 to 0.08]
  non-PT33F: number analyzed (Participants) | 42 | 40
  non-PT33F | 0.88 [0.57 to 1.34] | 0.06 [0.04 to 0.08]
Statistical Analysis 1: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT1 GMC Ratio (V114/Prevnar 13®); PT1 GMC Ratio = 0.52, 95% CI 2-sided [0.39 to 0.70]
Statistical Analysis 2: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT3 GMC Ratio (V114/Prevnar 13®); PT3 GMC Ratio = 1.79, 95% CI 2-sided [1.33 to 2.41]
Statistical Analysis 3: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT4 GMC Ratio (V114/Prevnar 13®); PT4 GMG Ratio = 0.87, 95% CI 2-sided [0.65 to 1.16]
Statistical Analysis 4: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT5 GMC Ratio (V114/Prevnar 13®); PT5 GMC Ratio = 0.51, 95% CI 2-sided [0.35 to 0.74]
Statistical Analysis 5: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT6A GMC Ratio (V114/Prevnar 13®); PT6A GMC Ratio = 0.31, 95% CI 2-sided [0.17 to 0.58]
Statistical Analysis 6: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT6B GMC Ratio (V114/Prevnar 13®); PT6B GMG Ratio = 0.16, 95% CI 2-sided [0.08 to 0.34]
Statistical Analysis 7: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT7F GMC Ratio (V114/Prevnar 13®); PT7F GMC Ratio = 0.48, 95% CI 2-sided [0.34 to 0.67]
Statistical Analysis 8: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT9V GMC Ratio (V114/Prevnar 13®); PT9V GMC Ratio = 0.56, 95% CI 2-sided [0.39 to 0.82]
Statistical Analysis 9: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT14 GMC Ratio (V114/Prevnar®); PT9V GMC Ratio = 0.64, 95% CI 2-sided [0.42 to 0.97]
Statistical Analysis 10: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT18C GMC Ratio (V114/Prevnar 13®); PT18C GMC Ratio = 0.85, 95% CI 2-sided [0.60 to 1.21]
Statistical Analysis 11: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT19A GMC Ratio (V114/Prevnar 13®); PT19A GMC Ratio = 0.66, 95% CI 2-sided [0.46 to 0.95]
Statistical Analysis 12: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT19F GMC Ratio (V114/Prevnar 13®); PT19F GMC Ratio = 1.11, 95% CI 2-sided [0.77 to 1.60]
Statistical Analysis 13: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT23F GMC Ratio (V114/Prevnar 13®); PT23F GMC Ratio = 0.68, 95% CI 2-sided [0.43 to 1.07]
Statistical Analysis 14: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — non-PT22F GMC Ratio (V114/Prevnar 13®); non-PT22F GMC Ratio = 44.61, 95% CI 2-sided [30.42 to 65.43]
Statistical Analysis 15: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — non-PT33F GMC Ratio (V114/Prevnar 13®); non-PT33F GMC Ratio = 15.29, 95% CI 2-sided [8.58 to 27.26]

7. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibodies at 1 Month Postdose 3 (PD3) in Infants: V114 2x:2x:2x vs. Prevnar 13®
Description: as for outcome 5
Time Frame: Month 7 (1 month PD3)
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Infant V114: 2x:2x:2x: Infants receive 4 total V114: 2x:2x:2x (containing 4.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 μg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
Arm/Group | Infant V114: 2x:2x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51
µg/mL
  PT1: number analyzed (Participants) | 33 | 40
  PT1 | 1.16 [0.94 to 1.42] | 1.48 [1.20 to 1.83]
  PT3: number analyzed (Participants) | 33 | 40
  PT3 | 1.15 [0.95 to 1.41] | 0.43 [0.35 to 0.54]
  PT4: number analyzed (Participants) | 33 | 40
  PT4 | 1.48 [1.17 to 1.87] | 0.98 [0.78 to 1.22]
  PT5: number analyzed (Participants) | 33 | 40
  PT5 | 1.11 [0.82 to 1.50] | 1.63 [1.25 to 2.14]
  PT6A: number analyzed (Participants) | 33 | 39
  PT6A | 0.91 [0.50 to 1.67] | 2.75 [2.28 to 3.31]
  PT6B: number analyzed (Participants) | 33 | 40
  PT6B | 0.24 [0.13 to 0.44] | 2.24 [1.54 to 3.24]
  PT7F: number analyzed (Participants) | 33 | 40
  PT7F | 2.12 [1.54 to 2.91] | 2.90 [2.48 to 3.39]
  PT9V: number analyzed (Participants) | 33 | 40
  PT9V | 1.18 [0.87 to 1.61] | 1.35 [1.05 to 1.74]
  PT14: number analyzed (Participants) | 33 | 40
  PT14 | 5.17 [3.83 to 6.99] | 5.01 [3.94 to 6.38]
  PT18C: number analyzed (Participants) | 33 | 40
  PT18C | 1.35 [0.97 to 1.88] | 1.41 [1.14 to 1.74]
  PT19A: number analyzed (Participants) | 33 | 40
  PT19A | 1.37 [0.94 to 1.99] | 1.45 [1.13 to 1.86]
  PT19F: number analyzed (Participants) | 33 | 40
  PT19F | 2.35 [1.59 to 3.47] | 1.89 [1.56 to 2.30]
  PT23F: number analyzed (Participants) | 33 | 40
  PT23F | 0.85 [0.55 to 1.31] | 1.13 [0.87 to 1.47]
  non-PT22F: number analyzed (Participants) | 33 | 40
  non-PT22F | 4.72 [3.46 to 6.43] | 0.06 [0.05 to 0.08]
  non-PT33F: number analyzed (Participants) | 33 | 40
  non-PT33F | 0.90 [0.51 to 1.57] | 0.06 [0.04 to 0.08]
Statistical Analysis 1: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT1 GMC Ratio (V114/Prevnar 13®); PT1 GMC Ratio = 0.78, 95% CI 2-sided [0.57 to 1.07]
Statistical Analysis 2: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT3 GMC Ratio (V114/Prevnar 13®); PT3 GMC Ratio = 2.68, 95% CI 2-sided [1.95 to 3.68]
Statistical Analysis 3: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT4 GMC Ratio (V114/Prevnar 13®); PT4 GMG Ratio = 1.52, 95% CI 2-sided [1.11 to 2.07]
Statistical Analysis 4: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT5 GMC Ratio (V114/Prevnar 13®); PT5 GMC Ratio = 0.68, 95% CI 2-sided [0.46 to 1.02]
Statistical Analysis 5: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT6A GMC Ratio (V114/Prevnar 13®); PT6A GMC Ratio = 0.33, 95% CI 2-sided [0.17 to 0.64]
Statistical Analysis 6: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT6B GMC Ratio (V114/Prevnar 13®); PT6B GMG Ratio = 0.11, 95% CI 2-sided [0.05 to 0.23]
Statistical Analysis 7: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT7F GMC Ratio (V114/Prevnar 13®); PT7F GMC Ratio = 0.73, 95% CI 2-sided [0.51 to 1.04]
Statistical Analysis 8: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT9V GMC Ratio (V114/Prevnar 13®); PT9V GMC Ratio = 0.88, 95% CI 2-sided [0.59 to 1.30]
Statistical Analysis 9: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT14 GMC Ratio (V114/Prevnar®); PT9V GMC Ratio = 1.03, 95% CI 2-sided [0.66 to 1.60]
Statistical Analysis 10: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT18C GMC Ratio (V114/Prevnar 13®); PT18C GMC Ratio = 0.96, 95% CI 2-sided [0.66 to 1.39]
Statistical Analysis 11: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT19A GMC Ratio (V114/Prevnar 13®); PT19A GMC Ratio = 0.95, 95% CI 2-sided [0.64 to 1.39]
Statistical Analysis 12: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT19F GMC Ratio (V114/Prevnar 13®); PT19F GMC Ratio = 1.24, 95% CI 2-sided [0.84 to 1.84]
Statistical Analysis 13: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT23F GMC Ratio (V114/Prevnar 13®); PT23F GMC Ratio = 0.75, 95% CI 2-sided [0.46 to 1.23]
Statistical Analysis 14: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — non-PT22F GMC Ratio (V114/Prevnar 13®); non-PT22F GMC Ratio = 77.57, 95% CI 2-sided [51.60 to 116.60]
Statistical Analysis 15: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — non-PT33F GMC Ratio (V114/Prevnar 13®); non-PT33F GMC Ratio = 15.66, 95% CI 2-sided [8.46 to 28.98]

8. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibodies at 1 Month Postdose 3 (PD3) in Infants: V114 0.5x:0.5x:2x vs. Prevnar 13®
Description: as for outcome 5
Time Frame: Month 7 (1 month PD3)
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Infant V114: 0.5x:0.5x:2x: Infants receive 4 total V114 0.5x:0.5x:2x (containing 1.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 2.0 μg of polysaccharide serotype 6B; and 250 μg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
Arm/Group | Infant V114: 0.5x:0.5x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 48 | 51
µg/mL
  PT1: number analyzed (Participants) | 37 | 40
  PT1 | 1.01 [0.79 to 1.29] | 1.48 [1.20 to 1.83]
  PT3: number analyzed (Participants) | 36 | 40
  PT3 | 0.95 [0.78 to 1.17] | 0.43 [0.35 to 0.54]
  PT4: number analyzed (Participants) | 36 | 40
  PT4 | 0.95 [0.78 to 1.19] | 0.98 [0.78 to 1.22]
  PT5: number analyzed (Participants) | 36 | 40
  PT5 | 0.87 [0.65 to 1.15] | 1.63 [1.25 to 2.14]
  PT6A: number analyzed (Participants) | 36 | 39
  PT6A | 1.35 [0.90 to 2.01] | 2.75 [2.28 to 3.31]
  PT6B: number analyzed (Participants) | 36 | 40
  PT6B | 0.80 [0.46 to 1.37] | 2.24 [1.54 to 3.24]
  PT7F: number analyzed (Participants) | 36 | 40
  PT7F | 1.73 [1.29 to 2.32] | 2.90 [2.48 to 3.39]
  PT9V: number analyzed (Participants) | 36 | 40
  PT9V | 1.07 [0.84 to 1.35] | 1.35 [1.05 to 1.74]
  PT14: number analyzed (Participants) | 37 | 40
  PT14 | 3.71 [2.67 to 5.17] | 5.01 [3.94 to 6.38]
  PT18C: number analyzed (Participants) | 37 | 40
  PT18C | 0.94 [0.69 to 1.27] | 1.41 [1.14 to 1.74]
  PT19A: number analyzed (Participants) | 37 | 40
  PT19A | 1.01 [0.80 to 1.28] | 1.45 [1.13 to 1.86]
  PT19F: number analyzed (Participants) | 37 | 40
  PT19F | 1.67 [1.35 to 2.07] | 1.89 [1.56 to 2.30]
  PT23F: number analyzed (Participants) | 36 | 40
  PT23F | 0.78 [0.61 to 1.00] | 1.13 [0.87 to 1.47]
  non-PT22F: number analyzed (Participants) | 36 | 40
  non-PT22F | 3.41 [2.74 to 4.25] | 0.06 [0.05 to 0.08]
  non-PT33F: number analyzed (Participants) | 37 | 40
  non-PT33F | 1.47 [0.97 to 2.23] | 0.06 [0.04 to 0.08]
Statistical Analysis 1: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT1 GMC Ratio (V114/Prevnar 13®); PT1 GMC Ratio = 0.68, 95% CI 2-sided [0.50 to 0.93]
Statistical Analysis 2: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT3 GMC Ratio (V114/Prevnar 13®); PT3 GMC Ratio = 2.21, 95% CI 2-sided [1.62 to 3.02]
Statistical Analysis 3: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT4 GMC Ratio (V114/Prevnar 13®); PT4 GMG Ratio = 0.97, 95% CI 2-sided [0.71 to 1.31]
Statistical Analysis 4: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT5 GMC Ratio (V114/Prevnar 13®); PT5 GMC Ratio = 0.53, 95% CI 2-sided [0.36 to 0.79]
Statistical Analysis 5: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT6A GMC Ratio (V114/Prevnar 13®); PT6A GMC Ratio = 0.49, 95% CI 2-sided [0.26 to 0.94]
Statistical Analysis 6: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT6B GMC Ratio (V114/Prevnar 13®); PT6B GMG Ratio = 0.36, 95% CI 2-sided [0.17 to 0.77]
Statistical Analysis 7: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT7F GMC Ratio (V114/Prevnar 13®); PT7F GMC Ratio = 0.60, 95% CI 2-sided [0.42 to 0.85]
Statistical Analysis 8: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT9V GMC Ratio (V114/Prevnar 13®); PT9V GMC Ratio = 0.79, 95% CI 2-sided [0.54 to 1.16]
Statistical Analysis 9: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT14 GMC Ratio (V114/Prevnar®); PT9V GMC Ratio = 0.74, 95% CI 2-sided [0.48 to 1.14]
Statistical Analysis 10: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT18C GMC Ratio (V114/Prevnar 13®); PT18C GMC Ratio = 0.66, 95% CI 2-sided [0.46 to 0.95]
Statistical Analysis 11: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT19A GMC Ratio (V114/Prevnar 13®); PT19A GMC Ratio = 0.70, 95% CI 2-sided [0.48 to 1.02]
Statistical Analysis 12: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT19F GMC Ratio (V114/Prevnar 13®); PT19F GMC Ratio = 0.88, 95% CI 2-sided [0.60 to 1.29]
Statistical Analysis 13: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT23F GMC Ratio (V114/Prevnar 13®); PT23F GMC Ratio = 0.69, 95% CI 2-sided [0.43 to 1.12]
Statistical Analysis 14: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — non-PT22F GMC Ratio (V114/Prevnar 13®); non-PT22F GMC Ratio = 56.08, 95% CI 2-sided [37.66 to 83.52]
Statistical Analysis 15: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — non-PT33F GMC Ratio (V114/Prevnar 13®); non-PT33F GMC Ratio = 25.75, 95% CI 2-sided [14.18 to 46.78]

9. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibodies at 1 Month Postdose 3 (PD3) in Infants: V114 1x:1x:2x vs. Prevnar 13®
Description: as for outcome 5
Time Frame: Month 7 (1 month PD3)
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Infant V114: 1x:1x:2x: Infants receive 4 total V114 1x:1x:2x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 250 μg of APA) total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
Arm/Group | Infant V114: 1x:1x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51
µg/mL
  PT1: number analyzed (Participants) | 34 | 40
  PT1 | 1.18 [0.94 to 1.49] | 1.48 [1.20 to 1.83]
  PT3: number analyzed (Participants) | 34 | 40
  PT3 | 1.10 [0.88 to 1.37] | 0.43 [0.35 to 0.54]
  PT4: number analyzed (Participants) | 34 | 40
  PT4 | 1.05 [0.81 to 1.35] | 0.98 [0.78 to 1.22]
  PT5: number analyzed (Participants) | 34 | 40
  PT5 | 0.83 [0.59 to 1.18] | 1.63 [1.25 to 2.14]
  PT6A: number analyzed (Participants) | 34 | 39
  PT6A | 0.92 [0.54 to 1.58] | 2.75 [2.28 to 3.31]
  PT6B: number analyzed (Participants) | 34 | 40
  PT6B | 0.39 [0.21 to 0.74] | 2.24 [1.54 to 3.24]
  PT7F: number analyzed (Participants) | 34 | 40
  PT7F | 1.71 [1.27 to 2.31] | 2.90 [2.48 to 3.39]
  PT9V: number analyzed (Participants) | 34 | 40
  PT9V | 0.92 [0.66 to 1.30] | 1.35 [1.05 to 1.74]
  PT14: number analyzed (Participants) | 34 | 40
  PT14 | 3.94 [3.02 to 5.14] | 5.01 [3.94 to 6.38]
  PT18C: number analyzed (Participants) | 34 | 40
  PT18C | 1.02 [0.77 to 1.35] | 1.41 [1.14 to 1.74]
  PT19A: number analyzed (Participants) | 34 | 40
  PT19A | 0.79 [0.58 to 1.08] | 1.45 [1.13 to 1.86]
  PT19F: number analyzed (Participants) | 37 | 40
  PT19F | 1.84 [1.35 to 2.52] | 1.89 [1.56 to 2.30]
  PT23F: number analyzed (Participants) | 36 | 40
  PT23F | 0.89 [0.58 to 1.38] | 1.13 [0.87 to 1.47]
  non-PT22F: number analyzed (Participants) | 36 | 40
  non-PT22F | 4.17 [3.10 to 5.62] | 0.06 [0.05 to 0.08]
  non-PT33F: number analyzed (Participants) | 37 | 40
  non-PT33F | 1.15 [0.71 to 1.86] | 0.06 [0.04 to 0.08]
Statistical Analysis 1: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT1 GMC Ratio (V114/Prevnar 13®); PT1 GMC Ratio = 0.80, 95% CI 2-sided [0.58 to 1.09]
Statistical Analysis 2: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT3 GMC Ratio (V114/Prevnar 13®); PT3 GMC Ratio = 2.55, 95% CI 2-sided [1.86 to 3.49]
Statistical Analysis 3: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT4 GMC Ratio (V114/Prevnar 13®); PT4 GMG Ratio = 1.07, 95% CI 2-sided [0.79 to 1.46]
Statistical Analysis 4: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT5 GMC Ratio (V114/Prevnar 13®); PT5 GMC Ratio = 0.51, 95% CI 2-sided [0.34 to 0.76]
Statistical Analysis 5: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT6A GMC Ratio (V114/Prevnar 13®); PT6A GMC Ratio = 0.34, 95% CI 2-sided [0.17 to 0.65]
Statistical Analysis 6: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT6B GMC Ratio (V114/Prevnar 13®); PT6B GMG Ratio = 0.18, 95% CI 2-sided [0.08 to 0.38]
Statistical Analysis 7: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT7F GMC Ratio (V114/Prevnar 13®); PT7F GMC Ratio = 0.59, 95% CI 2-sided [0.41 to 0.84]
Statistical Analysis 8: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT9V GMC Ratio (V114/Prevnar 13®); PT9V GMC Ratio = 0.68, 95% CI 2-sided [0.46 to 1.01]
Statistical Analysis 9: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT14 GMC Ratio (V114/Prevnar®); PT9V GMC Ratio = 0.79, 95% CI 2-sided [0.51 to 1.22]
Statistical Analysis 10: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT18C GMC Ratio (V114/Prevnar 13®); PT18C GMC Ratio = 0.72, 95% CI 2-sided [0.50 to 1.05]
Statistical Analysis 11: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT19A GMC Ratio (V114/Prevnar 13®); PT19A GMC Ratio = 0.55, 95% CI 2-sided [0.37 to 0.80]
Statistical Analysis 12: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT19F GMC Ratio (V114/Prevnar 13®); PT19F GMC Ratio = 0.97, 95% CI 2-sided [0.66 to 1.44]
Statistical Analysis 13: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT23F GMC Ratio (V114/Prevnar 13®); PT23F GMC Ratio = 0.79, 95% CI 2-sided [0.49 to 1.28]
Statistical Analysis 14: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — non-PT22F GMC Ratio (V114/Prevnar 13®); non-PT22F GMC Ratio = 68.64, 95% CI 2-sided [45.81 to 102.84]
Statistical Analysis 15: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — non-PT33F GMC Ratio (V114/Prevnar 13®); non-PT33F GMC Ratio = 20.03, 95% CI 2-sided [10.88 to 36.88]

10. Primary Outcome: Estimated Fold-Rise Per-Unit Change in Serotype-specific Antibody Concentrations Following an Increase in Polysaccharide Concentrations in Infants at 1 Month Postdose 3 (PD3)
Description: A mulitvariate regression model was used to evaluate the impact of increasing polysaccharide concentration from 1x to 2x on the natural logarithm of serotype-specific antibody concentrations 1 month PD3. Data points show the mean estimated fold-rise-per-unit change in antibody concentration following an increase from 1x to 2x in polysaccharide concentration. For each Prevnar 13®-type (PT) or non-Prevnar 13®-type (non-PT) serotypes, values >1.0 show an increase in antibody concentration whereas values <1.0 show a decrease in antibody concentration.
Time Frame: Month 7 (1 month PD3)
Population: All randomized and treated infants with results available for the outcome measure and no protocol violations in the V114 arms are included. Results are pooled across arms to determine the impact of increased polysaccharide concentration on antibody concentrations across V114 formulations.
Measure: Mean (95% Confidence Interval); unit: Estimated Fold-rise per-unit Change
Groups:
- All Infant Participants: Infant participants in the V114 treatment arms are included.
Arm/Group | All Infant Participants
Number analyzed (Participants) | 249
Estimated Fold-rise per-unit Change
  PT1: number analyzed (Participants) | 184
  PT1 | 1.19 [1.00 to 1.42]
  PT3: number analyzed (Participants) | 183
  PT3 | 1.13 [0.94 to 1.35]
  PT4: number analyzed (Participants) | 183
  PT4 | 1.44 [1.22 to 1.69]
  PT5: number analyzed (Participants) | 183
  PT5 | 1.29 [1.07 to 1.55]
  PT6A: number analyzed (Participants) | 183
  PT6A | 1.09 [0.83 to 1.43]
  PT6B: number analyzed (Participants) | 183
  PT6B | 0.73 [0.51 to 1.05]
  PT7F: number analyzed (Participants) | 183
  PT7F | 1.40 [1.16 to 1.68]
  PT9V: number analyzed (Participants) | 183
  PT9V | 1.15 [0.95 to 1.38]
  PT14: number analyzed (Participants) | 184
  PT14 | 1.47 [1.13 to 1.91]
  PT18C: number analyzed (Participants) | 184
  PT18C | 1.45 [1.23 to 1.70]
  PT19A: number analyzed (Participants) | 184
  PT19A | 1.30 [1.09 to 1.54]
  PT19F: number analyzed (Participants) | 184
  PT19F | 1.47 [1.23 to 1.76]
  PT22F: number analyzed (Participants) | 183
  PT22F | 1.64 [1.32 to 2.04]
  non-PT23F: number analyzed (Participants) | 183
  non-PT23F | 1.20 [0.97 to 1.48]
  non-PT33F: number analyzed (Participants) | 184
  non-PT33F | 0.94 [0.69 to 1.27]

11. Secondary Outcome: Percentage of Infant Participants Achieving the Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Threshold Value of ≥0.35 μg/mL at 1 Month Postdose 3 (PD3): V114 Formulations With 2x Aluminum Phosphate Adjuvant (APA)
Description: The percentage of infant participants with antibody responses meeting the World Health Organization (WHO)-accepted threshold value of ≥0.35 μg/mL was determined for each Prevnar 13®-type (PT) or non-Prevnar 13®-type (non-PT) pneumococcal serotype. Antibody levels were determined with the pneumococcal electrochemiluminescence (Pn ECL) assay for each V114 formulation with 2x APA and varying pneumococcal polysaccharide.
Time Frame: Month 7 (1 month PD3)
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Infant V114: 0.5x:0.5x:2x: Infants receive 4 total V114: 1x:1x:1x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 125 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
Arm/Group | Infant V114: 0.5x:0.5x:2x | Infant V114: 2x:1x:2x | Infant V114: 2x:2x:2x | Infant V114: 1x:1x:2x
Number analyzed (Participants) | 48 | 51 | 50 | 50
Percentage of Participants
  PT1: number analyzed (Participants) | 37 | 42 | 33 | 34
  PT1 | 94.6 [81.81 to 99.34] | 85.7 [71.46 to 94.57] | 97.0 [84.24 to 99.92] | 97.1 [84.67 to 99.93]
  PT3: number analyzed (Participants) | 36 | 42 | 33 | 34
  PT3 | 91.7 [77.53 to 98.25] | 85.7 [71.46 to 94.57] | 100.0 [89.42 to 100.00] | 88.2 [72.55 to 96.70]
  PT4: number analyzed (Participants) | 36 | 42 | 33 | 34
  PT4 | 91.7 [77.53 to 98.25] | 95.2 [83.84 to 99.42] | 97.0 [84.24 to 99.92] | 88.2 [72.55 to 96.70]
  PT5: number analyzed (Participants) | 36 | 42 | 33 | 34
  PT5 | 88.9 [73.94 to 96.89] | 78.6 [63.19 to 89.70] | 93.9 [79.77 to 99.26] | 88.2 [72.55 to 96.70]
  PT6A: number analyzed (Participants) | 36 | 42 | 33 | 34
  PT6A | 91.7 [77.53 to 98.25] | 66.7 [50.45 to 80.43] | 72.7 [54.48 to 86.70] | 76.5 [58.83 to 89.25]
  PT6B: number analyzed (Participants) | 36 | 42 | 33 | 34
  PT6B | 69.4 [51.89 to 83.65] | 47.6 [32.00 to 63.58] | 33.3 [17.96 to 51.83] | 52.9 [35.13 to 70.22]
  PT7F: number analyzed (Participants) | 36 | 42 | 33 | 34
  PT7F | 97.2 [85.47 to 99.93] | 100.00 [91.59 to 100.00] | 93.9 [79.77 to 99.26] | 97.1 [84.67 to 99.93]
  PT9V: number analyzed (Participants) | 36 | 42 | 33 | 34
  PT9V | 94.4 [81.34 to 99.32] | 78.6 [63.19 to 89.70] | 87.9 [71.80 to 96.60] | 85.3 [68.94 to 95.05]
  PT14: number analyzed (Participants) | 37 | 42 | 33 | 34
  PT14 | 94.6 [81.81 to 99.34] | 97.6 [87.43 to 99.94] | 100.00 [89.42 to 100.0] | 100.0 [89.72 to 100.00]
  PT18C: number analyzed (Participants) | 37 | 42 | 33 | 34
  PT18C | 91.9 [78.09 to 98.30] | 90.5 [77.38 to 97.34] | 93.9 [79.77 to 99.26] | 94.1 [80.32 to 99.28]
  PT19A: number analyzed (Participants) | 37 | 42 | 33 | 34
  PT19A | 91.9 [78.09 to 98.30] | 88.1 [74.37 to 96.02] | 93.9 [79.77 to 99.26] | 88.2 [72.55 to 96.70]
  PT19F: number analyzed (Participants) | 37 | 42 | 33 | 34
  PT19F | 97.3 [85.84 to 99.93] | 95.2 [83.84 to 99.42] | 97.0 [84.24 to 99.92] | 94.1 [80.32 to 99.28]
  PT23F: number analyzed (Participants) | 36 | 42 | 33 | 34
  PT23F | 83.3 [67.19 to 93.63] | 78.6 [63.19 to 89.70] | 84.8 [68.10 to 94.89] | 85.3 [68.94 to 95.05]
  non-PT22F: number analyzed (Participants) | 36 | 42 | 33 | 34
  non-PT22F | 100.00 [90.26 to 100.0] | 97.6 [87.43 to 99.94] | 97.0 [84.24 to 99.92] | 100.0 [89.72 to 100.00]
  non-PT33F: number analyzed (Participants) | 37 | 42 | 33 | 34
  non-PT33F | 91.9 [78.09 to 98.30] | 76.2 [60.55 to 87.95] | 72.7 [54.48 to 86.70] | 82.4 [65.47 to 93.24]

12. Secondary Outcome: Percentage of Infant Participants Achieving the Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Threshold Value of ≥0.35 μg/mL at 1 Month Postdose 3 (PD3): V114 Formulations With 1x Aluminum Phosphate Adjuvant (APA)
Description: The percentage of infant participants with antibody responses meeting the World Health Organization (WHO)-accepted threshold value of ≥0.35 μg/mL was determined for each Prevnar 13®-type (PT) or non-Prevnar 13®-type (non-PT) pneumococcal serotype. Antibody levels were determined with the pneumococcal electrochemiluminescence (Pn ECL) assay for each V114 formulation with 1x APA and varying pneumococcal polysaccharide.
Time Frame: Month 7 (1 month PD3)
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Infant V114: 1x:1x:1x
Number analyzed (Participants) | 50
Percentage of Participants
  PT1: number analyzed (Participants) | 38
  PT1 | 97.4 [86.19 to 99.93]
  PT3: number analyzed (Participants) | 38
  PT3 | 89.5 [75.20 to 97.06]
  PT4: number analyzed (Participants) | 38
  PT4 | 97.4 [86.19 to 99.93]
  PT5: number analyzed (Participants) | 38
  PT5 | 94.7 [82.25 to 99.36]
  PT6A: number analyzed (Participants) | 38
  PT6A | 86.8 [71.91 to 95.59]
  PT6B: number analyzed (Participants) | 38
  PT6B | 65.8 [48.65 to 80.37]
  PT7F: number analyzed (Participants) | 38
  PT7F | 100.0 [90.75 to 100.0]
  PT9V: number analyzed (Participants) | 38
  PT9V | 86.8 [71.91 to 95.59]
  PT14: number analyzed (Participants) | 38
  PT14 | 92.1 [78.62 to 98.34]
  PT18C: number analyzed (Participants) | 38
  PT18C | 97.4 [86.19 to 99.93]
  PT19A: number analyzed (Participants) | 38
  PT19A | 97.4 [86.19 to 99.93]
  PT19F: number analyzed (Participants) | 38
  PT19F | 100.0 [90.75 to 100.0]
  PT23F: number analyzed (Participants) | 38
  PT23F | 89.5 [75.20 to 97.06]
  non-PT22F: number analyzed (Participants) | 38
  non-PT22F | 94.7 [82.25 to 99.36]
  non-PT33F: number analyzed (Participants) | 38
  non-PT33F | 86.8 [71.91 to 95.59]

13. Secondary Outcome: Percentage of Infant Participants Achieving the Pneumococcal Immunoglobulin G (IgG) Serotype-specific Antibody Threshold Value of ≥0.35 μg/mL at 1 Month Postdose 4 (PD4): V114 1x:1x:1x vs Prenar 13®
Description: The percentage of infant participants with antibody responses meeting the World Health Organization (WHO)-accepted threshold value of ≥0.35 μg/mL was determined for each Prevnar 13®-type (PT) or non-Prevnar 13®-type (non-PT) pneumococcal serotype. Antibody levels were determined with the pneumococcal electrochemiluminescence (Pn ECL) assay for each V114 formulation.
Time Frame: One month following the 4th vaccination (approximately 13 to 16 months of age).
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infant V114: 1x:1x:1x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51
Percentage of Participants
  PT1: number analyzed (Participants) | 31 | 37
  PT1 | 96.8 | 100.0
  PT3: number analyzed (Participants) | 31 | 37
  PT3 | 90.3 | 75.7
  PT4: number analyzed (Participants) | 31 | 37
  PT4 | 90.3 | 97.3
  PT5: number analyzed (Participants) | 31 | 37
  PT5 | 100.0 | 100.0
  PT6A: number analyzed (Participants) | 31 | 37
  PT6A | 100.0 | 100.0
  PT6B: number analyzed (Participants) | 31 | 37
  PT6B | 100.0 | 100.0
  PT7F: number analyzed (Participants) | 31 | 37
  PT7F | 100.0 | 100.0
  PT9V: number analyzed (Participants) | 31 | 37
  PT9V | 100.0 | 100.0
  PT14: number analyzed (Participants) | 31 | 37
  PT14 | 100.0 | 100.0
  PT18C: number analyzed (Participants) | 31 | 37
  PT18C | 100.0 | 100.0
  PT19A: number analyzed (Participants) | 31 | 37
  PT19A | 100.0 | 100.0
  PT19F: number analyzed (Participants) | 31 | 37
  PT19F | 100.0 | 100.0
  PT23F: number analyzed (Participants) | 31 | 37
  PT23F | 100.0 | 100.0
  non-PT22F: number analyzed (Participants) | 31 | 37
  non-PT22F | 100.0 | 10.8
  non-PT33F: number analyzed (Participants) | 31 | 37
  non-PT33F | 100.0 | 2.7
Statistical Analysis 1: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT1 Percentage Point Difference (V114 - Prevnar 13®); PT1 Percentage Point Difference = -3.2, 95% CI 2-sided [-16.3 to 6.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT3 Percentage Point Difference (V114 - Prevnar 13®); PT3 Percentage Point Difference = 14.6, 95% CI 2-sided [-4.1 to 32.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT4 Percentage Point Difference (V114 - Prevnar 13®); PT4 Percentage Point Difference = -7.0, 95% CI 2-sided [-22.8 to 5.7] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT5 Percentage Point Difference (V114 - Prevnar 13®); PT5 Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT6A Percentage Point Difference (V114 - Prevnar 13®); PT6A Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 6: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT6B Percentage Point Difference (V114 - Prevnar 13®); PT6B Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 7: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT7F Percentage Point Difference (V114 - Prevnar 13®); PT7F Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 8: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT9V Percentage Point Difference (V114 - Prevnar 13®); PT9V Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 9: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT14 Percentage Point Difference (V114 - Prevnar 13®); PT14 Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 10: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT18C Percentage Point Difference (V114 - Prevnar 13®); PT18C Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 11: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT19A Percentage Point Difference (V114 - Prevnar 13®); PT19A Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 12: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT19F Percentage Point Difference (V114 - Prevnar 13®); PT19F Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 13: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — PT23F Percentage Point Difference (V114 - Prevnar 13®); PT23F Percentage Point Difference = 0.0, 95% CI 2-sided [-11.2 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 14: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — non-PT22F Percentage Point Difference (V114 - Prevnar 13®); non-PT22F Percentage Point Difference = 89.2, 95% CI 2-sided [75.2 to 95.7] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 15: Comparison: Infant V114: 1x:1x:1x vs Infant Prevnar 13®; Test type: Other — non-PT33F Percentage Point Difference (V114 - Prevnar 13®); non-PT33F Percentage Point Difference = 97.3, 95% CI 2-sided [85.1 to 99.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method

14. Secondary Outcome: Percentage of Infant Participants Achieving the Pneumococcal Immunoglobulin G (IgG) Serotype-specific Antibody Threshold Value of ≥0.35 μg/mL at 1 Month Postdose 4 (PD4): V114 2x:1x:2x vs Prenar 13®
Description: as for outcome 13
Time Frame: One month following the 4th vaccination (approximately 13 to 16 months of age).
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infant V114: 2x:1x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 51 | 51
Percentage of Participants
  PT1: number analyzed (Participants) | 24 | 37
  PT1 | 95.8 | 100.0
  PT3: number analyzed (Participants) | 24 | 37
  PT3 | 87.5 | 75.7
  PT4: number analyzed (Participants) | 23 | 37
  PT4 | 95.7 | 97.3
  PT5: number analyzed (Participants) | 24 | 37
  PT5 | 100.0 | 100.0
  PT6A: number analyzed (Participants) | 23 | 37
  PT6A | 100.0 | 100.0
  PT6B: number analyzed (Participants) | 23 | 37
  PT6B | 100.0 | 100.0
  PT7F: number analyzed (Participants) | 24 | 37
  PT7F | 100.0 | 100.0
  PT9V: number analyzed (Participants) | 24 | 37
  PT9V | 100.0 | 100.0
  PT14: number analyzed (Participants) | 24 | 37
  PT14 | 100.0 | 100.0
  PT18C: number analyzed (Participants) | 23 | 37
  PT18C | 100.0 | 100.0
  PT19A: number analyzed (Participants) | 24 | 37
  PT19A | 100.0 | 100.0
  PT19F: number analyzed (Participants) | 24 | 37
  PT19F | 100.0 | 100.0
  PT23F: number analyzed (Participants) | 24 | 37
  PT23F | 100.0 | 100.0
  non-PT22F: number analyzed (Participants) | 24 | 37
  non-PT22F | 95.8 | 10.8
  non-PT33F: number analyzed (Participants) | 23 | 37
  non-PT33F | 95.7 | 2.7
Statistical Analysis 1: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT1 Percentage Point Difference (V114 - Prevnar 13®); PT1 Percentage Point Difference = -4.2, 95% CI 2-sided [-20.4 to 5.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT3 Percentage Point Difference (V114 - Prevnar 13®); PT3 Percentage Point Difference = 11.8, 95% CI 2-sided [-10.0 to 30.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT4 Percentage Point Difference (V114 - Prevnar 13®); PT4 Percentage Point Difference = -1.6, 95% CI 2-sided [-18.8 to 10.3] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT5 Percentage Point Difference (V114 - Prevnar 13®); PT5 Percentage Point Difference = 0.0, 95% CI 2-sided [-14.0 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT6A Percentage Point Difference (V114 - Prevnar 13®); PT6A Percentage Point Difference = 0.0, 95% CI 2-sided [-14.5 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 6: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT6B Percentage Point Difference (V114 - Prevnar 13®); PT6B Percentage Point Difference = 0.0, 95% CI 2-sided [-14.5 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 7: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT7F Percentage Point Difference (V114 - Prevnar 13®); PT7F Percentage Point Difference = 0.0, 95% CI 2-sided [-14.0 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 8: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT9V Percentage Point Difference (V114 - Prevnar 13®); PT9V Percentage Point Difference = 0.0, 95% CI 2-sided [-14.0 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 9: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT14 Percentage Point Difference (V114 - Prevnar 13®); PT14 Percentage Point Difference = 0.0, 95% CI 2-sided [-14.0 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 10: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT18C Percentage Point Difference (V114 - Prevnar 13®); PT18C Percentage Point Difference = 0.0, 95% CI 2-sided [-14.5 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 11: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT19A Percentage Point Difference (V114 - Prevnar 13®); PT19A Percentage Point Difference = 0.0, 95% CI 2-sided [-14.0 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 12: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT19F Percentage Point Difference (V114 - Prevnar 13®); PT19F Percentage Point Difference = 0.0, 95% CI 2-sided [-14.0 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 13: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT23F Percentage Point Difference (V114 - Prevnar 13®); PT23F Percentage Point Difference = 0.0, 95% CI 2-sided [-14.0 to 9.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 14: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — non-PT22F Percentage Point Difference (V114 - Prevnar 13®); non-PT22F Percentage Point Difference = 85.0, 95% CI 2-sided [65.8 to 93.6] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 15: Comparison: Infant V114: 2x:1x:2x vs Infant Prevnar 13®; Test type: Other — non-PT33F Percentage Point Difference (V114 - Prevnar 13®); non-PT33F Percentage Point Difference = 92.9, 95% CI 2-sided [75.1 to 98.1] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method

15. Secondary Outcome: Percentage of Infant Participants Achieving the Pneumococcal Immunoglobulin G (IgG) Serotype-specific Antibody Threshold Value of ≥0.35 μg/mL at 1 Month Postdose 4 (PD4): V114 2x:2x:2x vs Prenar 13®
Description: as for outcome 13
Time Frame: One month following the 4th vaccination (approximately 13 to 16 months of age).
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infant V114: 2x:2x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51
Percentage of Participants
  PT1: number analyzed (Participants) | 33 | 37
  PT1 | 97.0 | 100.0
  PT3: number analyzed (Participants) | 33 | 37
  PT3 | 100.0 | 75.7
  PT4: number analyzed (Participants) | 33 | 37
  PT4 | 100.0 | 97.3
  PT5: number analyzed (Participants) | 33 | 37
  PT5 | 100.0 | 100.0
  PT6A: number analyzed (Participants) | 33 | 37
  PT6A | 100.0 | 100.0
  PT6B: number analyzed (Participants) | 33 | 37
  PT6B | 97.0 | 100.0
  PT7F: number analyzed (Participants) | 33 | 37
  PT7F | 100.0 | 100.0
  PT9V: number analyzed (Participants) | 33 | 37
  PT9V | 100.0 | 100.0
  PT14: number analyzed (Participants) | 33 | 37
  PT14 | 100.0 | 100.0
  PT18C: number analyzed (Participants) | 33 | 37
  PT18C | 100.0 | 100.0
  PT19A: number analyzed (Participants) | 33 | 37
  PT19A | 100.0 | 100.0
  PT19F: number analyzed (Participants) | 33 | 37
  PT19F | 100.0 | 100.0
  PT23F: number analyzed (Participants) | 33 | 37
  PT23F | 97.0 | 100.0
  non-PT22F: number analyzed (Participants) | 33 | 37
  non-PT22F | 100.0 | 10.8
  non-PT33F: number analyzed (Participants) | 33 | 37
  non-PT33F | 100.0 | 2.7
Statistical Analysis 1: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT1 Percentage Point Difference (V114 - Prevnar 13®); PT1 Percentage Point Difference = -3.0, 95% CI 2-sided [-15.5 to 6.7] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT3 Percentage Point Difference (V114 - Prevnar 13®); PT3 Percentage Point Difference = 24.3, 95% CI 2-sided [12.6 to 40.2] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT4 Percentage Point Difference (V114 - Prevnar 13®); PT4 Percentage Point Difference = 2.7, 95% CI 2-sided [-8.0 to 14.0] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT5 Percentage Point Difference (V114 - Prevnar 13®); PT5 Percentage Point Difference = 0.0, 95% CI 2-sided [-10.6 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT6A Percentage Point Difference (V114 - Prevnar 13®); PT6A Percentage Point Difference = 0.0, 95% CI 2-sided [-10.6 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 6: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT6B Percentage Point Difference (V114 - Prevnar 13®); PT6B Percentage Point Difference = -3.0, 95% CI 2-sided [-15.5 to 6.7] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 7: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT7F Percentage Point Difference (V114 - Prevnar 13®); PT7F Percentage Point Difference = 0.0, 95% CI 2-sided [-10.6 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 8: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT9V Percentage Point Difference (V114 - Prevnar 13®); PT9V Percentage Point Difference = 0.0, 95% CI 2-sided [-10.6 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 9: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT14 Percentage Point Difference (V114 - Prevnar 13®); PT14 Percentage Point Difference = 0.0, 95% CI 2-sided [-10.6 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 10: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT18C Percentage Point Difference (V114 - Prevnar 13®); PT18C Percentage Point Difference = 0.0, 95% CI 2-sided [-10.6 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 11: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT19A Percentage Point Difference (V114 - Prevnar 13®); PT19A Percentage Point Difference = 0.0, 95% CI 2-sided [-10.6 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 12: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT19F Percentage Point Difference (V114 - Prevnar 13®); PT19F Percentage Point Difference = 0.0, 95% CI 2-sided [-10.6 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 13: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — PT23F Percentage Point Difference (V114 - Prevnar 13®); PT23F Percentage Point Difference = -3.0, 95% CI 2-sided [-15.5 to 6.7] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 14: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — non-PT22F Percentage Point Difference (V114 - Prevnar 13®); non-PT22F Percentage Point Difference = 89.2, 95% CI 2-sided [75.2 to 95.7] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 15: Comparison: Infant V114: 2x:2x:2x vs Infant Prevnar 13®; Test type: Other — non-PT33F Percentage Point Difference (V114 - Prevnar 13®); non-PT33F Percentage Point Difference = 97.3, 95% CI 2-sided [85.7 to 99.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method

16. Secondary Outcome: Percentage of Infant Participants Achieving the Pneumococcal Immunoglobulin G (IgG) Serotype-specific Antibody Threshold Value of ≥0.35 μg/mL at 1 Month Postdose 4 (PD4): V114 0.5x:0.5x:2x vs Prenar 13®
Description: as for outcome 13
Time Frame: One month following the 4th vaccination (approximately 13 to 16 months of age).
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infant V114: 0.5x:0.5x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 48 | 51
Percentage of Participants
  PT1: number analyzed (Participants) | 34 | 37
  PT1 | 100.0 | 100.0
  PT3: number analyzed (Participants) | 34 | 37
  PT3 | 94.1 | 75.7
  PT4: number analyzed (Participants) | 34 | 37
  PT4 | 82.4 | 97.3
  PT5: number analyzed (Participants) | 34 | 37
  PT5 | 100.0 | 100.0
  PT6A: number analyzed (Participants) | 34 | 37
  PT6A | 100.0 | 100.0
  PT6B: number analyzed (Participants) | 34 | 37
  PT6B | 100.0 | 100.0
  PT7F: number analyzed (Participants) | 34 | 37
  PT7F | 100.0 | 100.0
  PT9V: number analyzed (Participants) | 34 | 37
  PT9V | 100.0 | 100.0
  PT14: number analyzed (Participants) | 34 | 37
  PT14 | 100.0 | 100.0
  PT18C: number analyzed (Participants) | 34 | 37
  PT18C | 100.0 | 100.0
  PT19A: number analyzed (Participants) | 34 | 37
  PT19A | 100.0 | 100.0
  PT19F: number analyzed (Participants) | 34 | 37
  PT19F | 100.0 | 100.0
  PT23F: number analyzed (Participants) | 34 | 37
  PT23F | 94.1 | 100.0
  non-PT22F: number analyzed (Participants) | 34 | 37
  non-PT22F | 100.0 | 10.8
  non-PT33F: number analyzed (Participants) | 34 | 37
  non-PT33F | 100.0 | 2.7
Statistical Analysis 1: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT1 Percentage Point Difference (V114 - Prevnar 13®); PT1 Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT3 Percentage Point Difference (V114 - Prevnar 13®); PT3 Percentage Point Difference = 18.4, 95% CI 2-sided [1.7 to 35.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT4 Percentage Point Difference (V114 - Prevnar 13®); PT4 Percentage Point Difference = -14.9, 95% CI 2-sided [-31.4 to -1.2] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT5 Percentage Point Difference (V114 - Prevnar 13®); PT5 Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT6A Percentage Point Difference (V114 - Prevnar 13®); PT6A Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 6: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT6B Percentage Point Difference (V114 - Prevnar 13®); PT6B Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 7: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT7F Percentage Point Difference (V114 - Prevnar 13®); PT7F Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 8: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT9V Percentage Point Difference (V114 - Prevnar 13®); PT9V Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 9: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT14 Percentage Point Difference (V114 - Prevnar 13®); PT14 Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 10: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT18C Percentage Point Difference (V114 - Prevnar 13®); PT18C Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 11: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT19A Percentage Point Difference (V114 - Prevnar 13®); PT19A Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 12: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT19F Percentage Point Difference (V114 - Prevnar 13®); PT19F Percentage Point Difference = 0.0, 95% CI 2-sided [-10.3 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 13: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — PT23F Percentage Point Difference (V114 - Prevnar 13®); PT23F Percentage Point Difference = -5.9, 95% CI 2-sided [-19.2 to 3.9] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 14: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — non-PT22F Percentage Point Difference (V114 - Prevnar 13®); non-PT22F Percentage Point Difference = 89.2, 95% CI 2-sided [75.2 to 95.7] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 15: Comparison: Infant V114: 0.5x:0.5x:2x vs Infant Prevnar 13®; Test type: Other — non-PT33F Percentage Point Difference (V114 - Prevnar 13®); non-PT33F Percentage Point Difference = 97.3, 95% CI 2-sided [85.9 to 99.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method

17. Secondary Outcome: Percentage of Infant Participants Achieving the Pneumococcal Immunoglobulin G (IgG) Serotype-specific Antibody Threshold Value of ≥0.35 μg/mL at 1 Month Postdose 4 (PD4): V114 1x:1x:2x vs Prenar 13®
Description: as for outcome 13
Time Frame: One month following the 4th vaccination (approximately 13 to 16 months of age).
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infant V114: 1x:1x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51
Percentage of Participants
  PT1: number analyzed (Participants) | 29 | 37
  PT1 | 96.6 | 100.0
  PT3: number analyzed (Participants) | 29 | 37
  PT3 | 89.7 | 75.7
  PT4: number analyzed (Participants) | 29 | 37
  PT4 | 89.7 | 97.3
  PT5: number analyzed (Participants) | 29 | 37
  PT5 | 96.6 | 100.0
  PT6A: number analyzed (Participants) | 29 | 37
  PT6A | 100.0 | 100.0
  PT6B: number analyzed (Participants) | 29 | 37
  PT6B | 100.0 | 100.0
  PT7F: number analyzed (Participants) | 29 | 37
  PT7F | 100.0 | 100.0
  PT9V: number analyzed (Participants) | 29 | 37
  PT9V | 96.6 | 100.0
  PT14: number analyzed (Participants) | 29 | 37
  PT14 | 100.0 | 100.0
  PT18C: number analyzed (Participants) | 29 | 37
  PT18C | 96.6 | 100.0
  PT19A: number analyzed (Participants) | 29 | 37
  PT19A | 93.1 | 100.0
  PT19F: number analyzed (Participants) | 29 | 37
  PT19F | 96.6 | 100.0
  PT23F: number analyzed (Participants) | 29 | 37
  PT23F | 100.0 | 100.0
  non-PT22F: number analyzed (Participants) | 29 | 37
  non-PT22F | 100.0 | 10.8
  non-PT33F: number analyzed (Participants) | 29 | 37
  non-PT33F | 96.6 | 2.7
Statistical Analysis 1: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT1 Percentage Point Difference (V114 - Prevnar 13®); PT1 Percentage Point Difference = -3.4, 95% CI 2-sided [-17.3 to 6.3] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT3 Percentage Point Difference (V114 - Prevnar 13®); PT3 Percentage Point Difference = 14.0, 95% CI 2-sided [-5.5 to 32.0] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT4 Percentage Point Difference (V114 - Prevnar 13®); PT4 Percentage Point Difference = -7.6, 95% CI 2-sided [-24.2 to 5.2] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT5 Percentage Point Difference (V114 - Prevnar 13®); PT5 Percentage Point Difference = -3.4, 95% CI 2-sided [-17.3 to 6.3] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT6A Percentage Point Difference (V114 - Prevnar 13®); PT6A Percentage Point Difference = 0.0, 95% CI 2-sided [-11.9 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 6: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT6B Percentage Point Difference (V114 - Prevnar 13®); PT6B Percentage Point Difference = 0.0, 95% CI 2-sided [-11.9 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 7: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT7F Percentage Point Difference (V114 - Prevnar 13®); PT7F Percentage Point Difference = 0.0, 95% CI 2-sided [-11.9 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 8: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT9V Percentage Point Difference (V114 - Prevnar 13®); PT9V Percentage Point Difference = -3.4, 95% CI 2-sided [-17.3 to 6.3] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 9: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT14 Percentage Point Difference (V114 - Prevnar 13®); PT14 Percentage Point Difference = 0.0, 95% CI 2-sided [-11.9 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 10: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT18C Percentage Point Difference (V114 - Prevnar 13®); PT18C Percentage Point Difference = -3.4, 95% CI 2-sided [-17.3 to 6.3] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 11: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT19A Percentage Point Difference (V114 - Prevnar 13®); PT19A Percentage Point Difference = -6.9, 95% CI 2-sided [-22.1 to 3.0] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 12: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT19F Percentage Point Difference (V114 - Prevnar 13®); PT19F Percentage Point Difference = -3.4, 95% CI 2-sided [-17.3 to 6.3] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 13: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — PT23F Percentage Point Difference (V114 - Prevnar 13®); PT23F Percentage Point Difference = 0.0, 95% CI 2-sided [-11.9 to 9.5] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 14: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — non-PT22F Percentage Point Difference (V114 - Prevnar 13®); non-PT22F Percentage Point Difference = 89.2, 95% CI 2-sided [75.2 to 95.7] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method
Statistical Analysis 15: Comparison: Infant V114: 1x:1x:2x vs Infant Prevnar 13®; Test type: Other — non-PT33F Percentage Point Difference (V114 - Prevnar 13®); non-PT33F Percentage Point Difference = 93.8, 95% CI 2-sided [78.5 to 98.3] — Estimated difference and 95% CI are based on the Miettinen and Nurminen method

18. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibodies at 1 Month Postdose 4 (PD4) in Infants
Description: The IgG antibody GMCs of each Prevnar 13®-type (PT) or non-Prevnar 13® type (non-PT) serotype at 1 month PD4 following V114 or Prevnar 13® treatment were determined with the pneumococcal electrochemiluminescence (Pn ECL) assay.
Time Frame: One month following the 4th vaccination (approximately 13 to 16 months of age)
Population: Randomized and treated infants with results available for the outcome measure and no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infant V114: 1x:1x:1x | Infant V114: 2x:1x:2x | Infant V114: 2x:2x:2x | Infant V114: 0.5x:0.5x:2x | Infant V114: 1x:1x:2x | Infant Prevnar 13®
Number analyzed (Participants) | 50 | 51 | 50 | 48 | 50 | 51
µg/mL
  PT1: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT1 | 1.67 [1.16 to 2.41] | 1.85 [1.20 to 2.86] | 2.25 [1.79 to 2.82] | 1.62 [1.27 to 2.05] | 1.67 [1.22 to 2.28] | 2.33 [1.84 to 2.95]
  PT3: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT3 | 1.10 [0.81 to 1.51] | 0.96 [0.69 to 1.33] | 1.69 [1.40 to 2.03] | 1.06 [0.79 to 1.41] | 1.09 [0.77 to 1.52] | 0.62 [0.49 to 0.77]
  PT4: number analyzed (Participants) | 31 | 23 | 33 | 34 | 29 | 37
  PT4 | 1.71 [1.21 to 2.41] | 1.60 [1.07 to 2.39] | 2.46 [1.80 to 3.36] | 1.21 [0.82 to 1.78] | 1.39 [0.97 to 1.98] | 1.78 [1.33 to 2.39]
  PT5: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT5 | 2.31 [1.66 to 3.22] | 2.46 [1.76 to 3.43] | 3.61 [2.88 to 4.52] | 2.38 [1.72 to 3.30] | 2.50 [1.73 to 3.61] | 4.72 [3.80 to 5.86]
  PT6A: number analyzed (Participants) | 31 | 23 | 33 | 34 | 29 | 37
  PT6A | 6.93 [4.69 to 10.22] | 9.62 [6.96 to 13.31] | 6.16 [4.55 to 8.34] | 7.88 [5.84 to 10.64] | 6.58 [4.50 to 9.60] | 10.31 [8.22 to 12.92]
  PT6B: number analyzed (Participants) | 31 | 23 | 33 | 34 | 29 | 37
  PT6B | 7.35 [4.96 to 10.88] | 8.89 [5.87 to 13.46] | 6.31 [4.62 to 8.61] | 7.27 [5.40 to 9.77] | 6.53 [4.57 to 9.34] | 11.55 [9.30 to 14.35]
  PT7F: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT7F | 4.69 [3.44 to 6.40] | 3.00 [2.29 to 3.92] | 5.24 [3.94 to 6.99] | 4.65 [3.26 to 6.63] | 4.39 [3.33 to 5.79] | 5.65 [4.65 to 6.88]
  PT9V: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT9V | 2.96 [2.01 to 4.36] | 2.20 [1.56 to 3.10] | 3.18 [2.47 to 4.08] | 2.83 [2.08 to 3.84] | 2.27 [1.57 to 3.27] | 3.25 [2.47 to 4.29]
  PT14: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT14 | 8.68 [5.89 to 12.80] | 7.83 [5.48 to 11.20] | 9.40 [6.47 to 13.65] | 8.48 [6.28 to 11.45] | 7.15 [5.15 to 9.93] | 7.48 [5.79 to 9.67]
  PT18C: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT18C | 2.06 [1.54 to 2.77] | 2.82 [2.13 to 3.72] | 2.95 [2.32 to 3.75] | 2.21 [1.70 to 2.87] | 1.82 [1.30 to 2.56] | 2.84 [2.31 to 3.47]
  PT19A: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT19A | 3.65 [2.69 to 4.95] | 5.34 [3.79 to 7.53] | 6.54 [4.77 to 8.96] | 3.46 [2.48 to 4.81] | 5.86 [4.17 to 8.23] | 5.11 [4.19 to 6.23]
  PT19F: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT19F | 6.07 [4.40 to 8.37] | 9.72 [7.28 to 12.99] | 9.11 [7.00 to 11.84] | 4.38 [3.20 to 5.98] | 5.86 [4.17 to 8.23] | 5.11 [4.19 to 6.23]
  PT23F: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  PT23F | 2.01 [1.43 to 2.83] | 2.60 [1.84 to 3.67] | 2.95 [2.26 to 3.86] | 2.00 [1.36 to 2.94] | 2.02 [1.44 to 2.83] | 3.91 [3.03 to 5.05]
  non-PT22F: number analyzed (Participants) | 31 | 24 | 33 | 34 | 29 | 37
  non-PT22F | 7.21 [4.99 to 10.40] | 5.05 [3.13 to 8.14] | 10.66 [7.74 to 14.69] | 6.78 [5.06 to 9.09] | 7.88 [5.92 to 10.48] | 0.08 [0.06 to 0.12]
  non-PT33F: number analyzed (Participants) | 31 | 23 | 33 | 34 | 29 | 37
  non-PT33F | 6.44 [4.51 to 9.21] | 3.93 [2.24 to 6.88] | 8.03 [5.94 to 10.86] | 6.85 [4.98 to 9.42] | 5.07 [3.46 to 7.42] | 0.07 [0.05 to 0.09]

19. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibodies at 1 Month After Vaccination in Adults
Description: The IgG antibody GMCs of each Prevnar 13®-type (PT) or non-Prevnar 13® type (non-PT) serotype at 1 month after a single vaccination with V114 were determined with the pneumococcal electrochemiluminescence (Pn ECL) assay. Data reflect the GMC of each serotype.
Time Frame: Month 2 (1 month after a single vaccination)
Population: Randomized and treated adults with results available for the outcome measure and no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Adult V114: 1x:1x:1x | Adult V114: 2x.2x.2x
Number analyzed (Participants) | 20 | 20
µg/mL
  PT1: number analyzed (Participants) | 16 | 18
  PT1 | 3.19 [1.71 to 5.97] | 5.82 [3.34 to 10.15]
  PT3: number analyzed (Participants) | 16 | 18
  PT3 | 0.84 [0.47 to 1.47] | 1.12 [0.62 to 2.03]
  PT4: number analyzed (Participants) | 16 | 18
  PT4 | 2.28 [1.25 to 4.18] | 1.80 [1.08 to 2.99]
  PT5: number analyzed (Participants) | 16 | 18
  PT5 | 2.63 [1.01 to 6.84] | 1.90 [1.02 to 3.52]
  PT6A: number analyzed (Participants) | 16 | 18
  PT6A | 8.23 [4.26 to 15.86] | 3.52 [1.48 to 8.36]
  PT6B: number analyzed (Participants) | 16 | 18
  PT6B | 8.96 [4.15 to 19.34] | 4.08 [1.61 to 10.35]
  PT7F: number analyzed (Participants) | 16 | 18
  PT7F | 4.88 [2.22 to 10.75] | 2.20 [1.01 to 4.80]
  PT9V: number analyzed (Participants) | 16 | 18
  PT9V | 4.96 [2.33 to 10.56] | 2.96 [1.70 to 5.15]
  PT14: number analyzed (Participants) | 16 | 18
  PT14 | 16.24 [7.42 to 35.54] | 18.45 [7.56 to 45.02]
  PT18C: number analyzed (Participants) | 16 | 18
  PT18C | 4.56 [2.32 to 8.98] | 2.63 [1.52 to 4.56]
  PT19A: number analyzed (Participants) | 16 | 18
  PT19A | 9.71 [4.98 to 18.94] | 4.39 [2.29 to 8.42]
  PT19F: number analyzed (Participants) | 16 | 18
  PT19F | 3.39 [1.61 to 7.15] | 3.71 [1.70 to 8.09]
  PT22F: number analyzed (Participants) | 16 | 18
  PT22F | 6.05 [2.66 to 13.75] | 7.81 [3.84 to 15.87]
  non-PT23F: number analyzed (Participants) | 16 | 18
  non-PT23F | 4.78 [2.03 to 11.26] | 3.32 [1.49 to 7.38]
  non-PT33F: number analyzed (Participants) | 16 | 18
  non-PT33F | 3.41 [1.64 to 7.08] | 4.69 [1.51 to 14.53]

20. Secondary Outcome: Percentage of Participants With ≥4-fold-rise From Baseline in Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibodies at 1 Month After Vaccination in Adults
Description: The percentage of participants with ≥4-fold-rise from baseline in each Prevnar 13®-type (PT) or non-Prevnar 13® type (non-PT) serotype at 1 month after a single vaccination with V114 were determined with the pneumococcal electrochemiluminescence (Pn ECL) assay.
Time Frame: Month 2 (1 month after a single vaccination)
Population: Randomized and treated adults with results available for the outcome measure and no protocol violations are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Adult V114: 1x:1x:1x | Adult V114: 2x.2x.2x
Number analyzed (Participants) | 20 | 20
Percentage of Participants
  PT1: number analyzed (Participants) | 16 | 18
  PT1 | 93.75 [69.77 to 99.84] | 100.00 [81.47 to 100.00]
  PT3: number analyzed (Participants) | 16 | 18
  PT3 | 56.25 [29.88 to 80.25] | 66.67 [40.99 to 86.66]
  PT4: number analyzed (Participants) | 16 | 18
  PT4 | 93.75 [69.77 to 99.84] | 88.89 [65.29 to 98.62]
  PT5: number analyzed (Participants) | 16 | 18
  PT5 | 50.00 [24.65 to 75.35] | 61.11 [35.75 to 82.70]
  PT6A: number analyzed (Participants) | 16 | 18
  PT6A | 81.25 [54.35 to 95.95] | 72.22 [46.52 to 90.31]
  PT6B: number analyzed (Participants) | 16 | 18
  PT6B | 100.00 [79.41 to 100.0] | 83.33 [58.58 to 96.42]
  PT7F: number analyzed (Participants) | 16 | 18
  PT7F | 81.25 [54.35 to 95.95] | 44.44 [21.53 to 69.24]
  PT9V: number analyzed (Participants) | 16 | 18
  PT9V | 100.00 [79.41 to 100.00] | 88.89 [65.29 to 98.62]
  PT14: number analyzed (Participants) | 16 | 18
  PT14 | 87.50 [61.65 to 98.45] | 83.33 [58.58 to 96.42]
  PT18C: number analyzed (Participants) | 16 | 18
  PT18C | 87.50 [61.65 to 98.45] | 72.22 [46.52 to 90.31]
  PT19A: number analyzed (Participants) | 16 | 18
  PT19A | 81.25 [54.35 to 95.95] | 55.56 [30.76 to 78.47]
  PT19F: number analyzed (Participants) | 16 | 18
  PT19F | 81.25 [54.35 to 95.95] | 83.33 [58.58 to 96.42]
  PT22F: number analyzed (Participants) | 16 | 18
  PT22F | 93.75 [69.77 to 99.84] | 83.33 [58.58 to 96.42]
  non-PT23F: number analyzed (Participants) | 16 | 18
  non-PT23F | 87.50 [61.65 to 98.45] | 77.78 [52.36 to 93.59]
  non-PT33F: number analyzed (Participants) | 16 | 18
  non-PT33F | 62.50 [35.43 to 84.80] | 66.67 [40.99 to 86.66]

21. Primary Outcome: Estimated Fold-Rise Per-Unit Change on Serotype-specific Antibody Concentrations Following an Increase in Aluminum Phosphate Adjuvant (APA) Concentration 1 Month Postdose 3 (PD3) in Infants
Description: A mulitvariate regression model was used to evaluate the impact of increasing APA concentration on the natural logarithm of serotype-specific antibody concentrations 1 month PD3. Data points show the mean estimated fold-rise-per-unit change in antibody concentration following an increase in APA. For each Prevnar 13®-type (PT) or non-Prevnar 13®-type (non-PT) serotypes, values >1.0 show an increase in antibody concentration whereas values <1.0 show a decrease in antibody concentration.
Time Frame: Month 7 (1 month PD3)
Population: All randomized and treated infants with results available for the outcome measure and no protocol violations in the V114 arms are included.
Measure: Mean (95% Confidence Interval); unit: Estimated Fold-rise per-unit Change
Groups:
- All V114 Infant Participants: All infant participants in the V114 treatment arms are included.
Arm/Group | All V114 Infant Participants
Number analyzed (Participants) | 249
Estimated Fold-rise per-unit Change
  PT1: number analyzed (Participants) | 184
  PT1 | 0.84 [0.68 to 1.03]
  PT3: number analyzed (Participants) | 183
  PT3 | 0.84 [0.68 to 1.04]
  PT4: number analyzed (Participants) | 183
  PT4 | 0.77 [0.63 to 0.95]
  PT5: number analyzed (Participants) | 183
  PT5 | 0.76 [0.61 to 0.95]
  PT6A: number analyzed (Participants) | 183
  PT6A | 0.89 [0.66 to 1.20]
  PT6B: number analyzed (Participants) | 183
  PT6B | 0.74 [0.52 to 1.05]
  PT7F: number analyzed (Participants) | 183
  PT7F | 1.01 [0.81 to 1.26]
  PT9V: number analyzed (Participants) | 183
  PT9V | 0.83 [0.66 to 1.04]
  PT14: number analyzed (Participants) | 184
  PT14 | 1.48 [1.16 to 1.89]
  PT18C: number analyzed (Participants) | 184
  PT18C | 0.75 [0.60 to 0.94]
  PT19A: number analyzed (Participants) | 184
  PT19A | 0.77 [0.61 to 0.97]
  PT19F: number analyzed (Participants) | 184
  PT19F | 1.01 [0.79 to 1.27]
  PT22F: number analyzed (Participants) | 183
  PT22F | 1.37 [1.09 to 1.73]
  non-PT23F: number analyzed (Participants) | 183
  non-PT23F | 0.73 [0.57 to 0.95]
  non-PT33F: number analyzed (Participants) | 184
  non-PT33F | 1.00 [0.75 to 1.33]

ADVERSE EVENTS:
Time Frame: Up to 14 days after each dose of study drug.
Description: All adult and infant participants who received ≥1 dose of study drug are included.
Groups:
- Adult: V114-1x:1x:1x: On Day 1, adults receive a single vaccination of V114 1x:1x:1x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 125 µg of APA).
- Adult: V114-2x:2x:2x: On Day 1, adults receive a single vaccination of V114 2x:2x:2x (containing 4.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 µg of APA).
- Infant: V114-1x:1x:1x: Infants receive 4 total V114: 1x:1x:1x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 125 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant: V114-2x:1x:2x: Infants receive 4 total V114: 2x:1x:2x (containing 4.0 μg of polysaccharide serotypes 6A, 18C, 19A, 19F, and 23F; 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 7F, 9V, 14, 22F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant: V114-2x:2x:2x: Infants receive 4 total V114: 2x:2x:2x (containing 4.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 8.0 μg of polysaccharide serotype 6B; and 250 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant: V114-0.5x:0.5x:2x: Infants receive 4 total V114 0.5x:0.5x:2x (containing 1.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 2.0 μg of polysaccharide serotype 6B; and 250 µg of APA) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant: V114-1x:1x:2x: Infants receive 4 total V114 1x:1x:2x (containing 2.0 μg of polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; 4.0 μg of polysaccharide serotype 6B; and 250 µg of APA) total vaccinations given at 2, 4, 6, and 12 to 15 months of age.
- Infant: Prevnar 13: Infants receive 4 total Prevnar 13® (containing 2.2 µg of pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, and 23F; and 4.4 µg of serotype 6B) vaccinations given at 2, 4, 6, and 12 to 15 months of age.
Arm/Group | Adult: V114-1x:1x:1x | Adult: V114-2x:2x:2x | Infant: V114-1x:1x:1x | Infant: V114-2x:1x:2x | Infant: V114-2x:2x:2x | Infant: V114-0.5x:0.5x:2x | Infant: V114-1x:1x:2x | Infant: Prevnar 13
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/50 | 0/51 | 0/50 | 0/48 | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/50 | 4/51 | 3/50 | 3/48 | 0/50 | 5/51
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20 | 49/50 | 51/51 | 48/50 | 46/48 | 49/50 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult: V114-1x:1x:1x (N=20) | Adult: V114-2x:2x:2x (N=20) | Infant: V114-1x:1x:1x (N=50) | Infant: V114-2x:1x:2x (N=51) | Infant: V114-2x:2x:2x (N=50) | Infant: V114-0.5x:0.5x:2x (N=48) | Infant: V114-1x:1x:2x (N=50) | Infant: Prevnar 13 (N=51)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult: V114-1x:1x:1x (N=20) | Adult: V114-2x:2x:2x (N=20) | Infant: V114-1x:1x:1x (N=50) | Infant: V114-2x:1x:2x (N=51) | Infant: V114-2x:2x:2x (N=50) | Infant: V114-0.5x:0.5x:2x (N=48) | Infant: V114-1x:1x:2x (N=50) | Infant: Prevnar 13 (N=51)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Plagiocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (8) | 4 (9) | 4 (4) | 6 (7) | 6 (8) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 4 (4) | 0 (0) | 0 (0) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infantile spitting up (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 3 (3) | 5 (9) | 1 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (6) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (10) | 8 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 3 (4) | 3 (3)
Injection site erythema (General disorders) | 7 (8) | 6 (6) | 22 (48) | 33 (60) | 26 (51) | 29 (56) | 28 (47) | 27 (50)
Injection site granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 21 (37) | 27 (51) | 19 (36) | 26 (50) | 18 (33) | 14 (24)
Injection site joint pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site lymphadenopathy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site macule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 20 (25) | 20 (31) | 47 (104) | 46 (111) | 40 (114) | 37 (101) | 42 (94) | 41 (102)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 7 (7) | 6 (6) | 19 (36) | 28 (47) | 21 (30) | 25 (55) | 22 (42) | 20 (32)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 13 (15) | 16 (27) | 17 (31) | 13 (16) | 11 (14) | 13 (24)
Sluggishness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 2 (3)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 5 (5) | 7 (7) | 3 (4) | 2 (2) | 4 (5)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (3)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Roseola (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 7 (8) | 7 (7) | 9 (10) | 3 (3) | 5 (5)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stool pH decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 23 (60) | 31 (67) | 32 (73) | 27 (53) | 26 (53) | 27 (50)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lordosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 11 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Developmental coordination disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 9 (14) | 8 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 42 (137) | 43 (126) | 42 (120) | 36 (106) | 37 (101) | 37 (106)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 47 (186) | 49 (185) | 47 (189) | 40 (174) | 42 (151) | 47 (158)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stereotypy (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 5 (5) | 1 (2) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 6 (7) | 3 (4) | 2 (4) | 2 (2) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.